CLINICAL TRIAL: NCT06355518
Title: Pre-operative Immuno-nutrition in Patients Undergoing Radical Cystectomy for Bladder Cancer: a Multicentre, Randomised, Open-label, Parallel Group Study
Brief Title: Pre-operative Immuno-Nutrition in Radical Cystectomy
Acronym: INu-RC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INu-RC
Record Dates: First submitted 2024-03-19; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Immunonutrition Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative Immunonutrition (Experimental): Preoperative administration of a high-calorie, high-protein liquid oral nutritional supplement containing immunonutrients [Impact® Oral (237 mL per serving); Nestlé Health Science - Creully Sur Seulles - France]. Two units of Impact® Oral per day will be administered for 7 days before surgery.
  Interventions: Dietary Supplement: Immunonutrition
- Preoperative Standard Oral Nutritional Supplement (Active Comparator): Preoperative administration of a standard high-calorie-high-protein liquid oral nutritional supplement [Meritene® Protein Drink (200 mL per serving); Nestlé Health Science - Creully Sur Seulles - France]. Two units of Meritene® Protein Drink per day will be administered for 7 days before surgery.
  Interventions: Dietary Supplement: Standard Oral Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Immunonutrition — This formula is enriched in arginine, nucleotides (RNA) and omega-3 fatty acids and provides, with the proposed therapeutic volume (2 units per day), 36 grams of protein and 682 kcal/day.
  Other Names: Impact® Oral
  Arms: Preoperative Immunonutrition
Dietary Supplement: Standard Oral Nutritional Supplement — This formula provides 38 grams of protein and 500 kcal/day with the proposed therapeutic volume.
  Other Names: Meritene® Drink
  Arms: Preoperative Standard Oral Nutritional Supplement

SUMMARY:
This study will evaluate the effect of preoperative oral immunonutrition on postoperative complications in patients undergoing radical cystectomy for bladder cancer. Patients receiving preoperative immunonutrition will be compared to controls receiving a standard high-calorie, high-protein oral nutritional supplement.

DETAILED DESCRIPTION:
Radical cystectomy with pelvic lymph node dissection and urinary reconstruction is a major surgical procedure performed for bladder cancer. The literature reports an incidence of 50-88% and 30-42% for any grade complications (Clavier-Dindo grade I-IV) and severe complications (Clavier-Dindo grade ≥III), respectively. Nutritional status prior to radical cystectomy has been shown to be a strong predictor of 90-day mortality. The term "immunonutrition" refers to the oral or enteral administration of specific substrates such as omega-3 fatty acids, arginine, and nucleotides. These substrates have been shown to upregulate the host immune response, modulate inflammatory responses and improve protein synthesis after surgery, with a favorable impact on postoperative infection rates and length of hospital stay in major abdominal surgery. Data on patients undergoing radical cystectomy are scarce, mainly due to the small sample size of the studies. However, the available evidence suggests a potential beneficial effect of this nutritional intervention in patients undergoing radical cystectomy. Several aspects remain largely unclear, including the dosage and timing of immunonutrition and the impact of preoperative malnutrition risk on the efficacy of immunonutrition. This study will evaluate the effect of 7 days of preoperative immunonutrition on postoperative complications compared to patients receiving standard high-calorie, high-protein oral nutritional supplements.

ELIGIBILITY:
Inclusion Criteria:

* Surgical indication to radical cystectomy with diagnosis of muscle invasive bladder cancer (any N, any M), BCG (Bacillus Calmette-Guerin)-unresponsive non-muscle invasive bladder cancer or extensive non-muscle invasive bladder cancer that cannot be treated with endoscopic surgery alone;
* Willingness to participate by signing written informed consent.

Exclusion Criteria:

* Age < 18 years;
* Pregnant or lactating women;
* Participation in another study with nutritional supplements within the 30 days preceding and during the present study
* Known hypersensitivity or allergy to components of immunonutrition or standard high-calorie high-protein oral nutritional supplement;
* Need for artificial nutrition support due to totally compromised spontaneous food intake;
* Diarrhoea with suspected malabsorption syndrome;
* Inability to consume oral supplements as a consequence of pre-existing disease (e.g. dysphagia) or other factors (e.g. language barrier, psychological disorders, absence of a home caregiver in dependent or elderly patients);
* Kidney failure with need for renal replacement therapy;
* Type 1 diabetes mellitus;
* Type 2 diabetes mellitus requiring insulin therapy and/or inadequate glycaemic control (glycosylated haemoglobin ≥7% and/or fasting plasma glucose ≥150 mg/dL);
* Inability to give an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
30-day complications | 30 days after surgery
  Percentage of patients developing at least one post-operative complication (as detailed in the study protocol: infectious, urinary, gastrointestinal, and wound-related complications)

SECONDARY OUTCOMES:
30-day severe complications | 30 days after surgery
  Percentage of patients developing at least one Clavien-Dindo grade ≥III post-operative complication (as detailed in the study protocol: infectious, urinary, gastrointestinal, and wound-related complications)
90-day severe complications | 90 days after surgery
  Percentage of patients developing at least one Clavien-Dindo grade ≥III post-operative complication (as detailed in the study protocol: infectious, urinary, gastrointestinal, and wound-related complications)
30-day and 90-day infectious complications | 30 and 90 days after surgery
  Percentage of patients developing at least one infectious complication (as detailed in the study protocol)
30-day and 90-day occurrence of other medical conditions | 30 and 90 days after surgery
  Percentage of patients developing at least one other medical conditions (as detailed in the study protocol)
Time to recovery of bowel function | Immediately after surgery
  Time from surgery to first flatus counting the day of surgery as day 0
Time to postoperative mobilization | Immediately after surgery
  Time from surgery to first walk counting the day of surgery as day 0
Muscular strength modifications | Up hospital discharge, assessed up to 90 days
  Difference in hand-grip strength (mean of three consecutive measurements from dominant hand) and in the sit-and-stand test
Weight modifications | From preadmission visit to 90-day follow-up visit
  Difference in body weight
Biochemical nutritional indexes modifications | Up to hospital discharge, assessed up to 90 days
  Biochemical nutritional indexes
Need of blood transfusions | Immediately after surgery
  Percentage of patients undergoing blood transfusions (red blood cells, plasma, and/or platelets)
Length of stay | Immediately after surgery
  Time from hospital admission to discharge at home or to another facility
Readmission rate | 30 and 90 days after surgery
  Incidence of unplanned re-hospitalization due to all causes
30-day and 90-day mortality | 30 and 90 days after surgery
  Death rate due to all causes
Compliance | 7 days before surgery
  Percentage of patients consuming ≥80% of the prescribed supplement
Tolerability (gastrointestinal symptoms related to nutritional supplement) | 7 days before surgery
  Percentage of patients experiencing at least one moderate-severe adverse gastrointestinal effects

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casirati A, Da Prat V, Bettiga A, Aretano L, Trevisani F, Cereda E, Briganti A, Colombo E, Preziati G, De Simeis F, Salonia A, Montorsi F, Caccialanza R, Naspro R. Immunonutrition in Radical Cystectomy: State of the Art and Perspectives. Cancers (Basel). 2023 Jul 24;15(14):3747. doi: 10.3390/cancers15143747. PMID 37509408